CLINICAL TRIAL: NCT02268058
Title: The Use of Ibuprofen and Acetaminophen for Acute Headache in the Post Concussive Youth: A Pilot Study.
Brief Title: Use of Ibuprofen and Acetaminophen for Treatment of Acute Headache Post Concussion in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Dr.Tina Petrelli, McMaster Children's Hospital, McMaster Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NIF-Petrelli
Record Dates: First submitted 2014-10-09; First posted 2014-10-20 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Concussion; Headache
MeSH Terms: conditions — Brain Concussion; Headache | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- tx 1: acetaminophen and education (Active Comparator): Patient took routinely acetaminophen every 4 hours when awake for a 72 hour period and documented their headaches for a week.
  Patient and family received standard education on concussion management in the Emergency department.
  Interventions: Drug: Acetaminophen
- Tx 2: ibuprofen and education (Active Comparator): Patient took routinely ibuprofen every 6 hours when awake for a 72 hour period and documented their headaches for a week.
  Patient and family received standard education on concussion management in the Emergency department.
  Interventions: Drug: Ibuprofen
- Tx 3: ibuprofen/acetaminophen/education (Active Comparator): Patient took routinely ibuprofen (Q6H) and acetaminophen (Q4H) for when awake for 72 hours post concussion and documented their headaches for a week.
  Patient and family received standard education on concussion management in the Emergency Department.
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen
- Tx 4: no routine meds and education (No Intervention): Patient was advised to manage headaches as they typically would. There was no instruction given for the routine administration of either ibuprofen or acetaminophen.
  The Patient and family received standard education in the ER department and diarized their headaches and medications they took for a one week period.

INTERVENTIONS:
Drug: Acetaminophen — routine administration of medication for a 72 hour period
  Other Names: tylenol
  Arms: Tx 3: ibuprofen/acetaminophen/education; tx 1: acetaminophen and education
Drug: Ibuprofen — routine administration of medication for a 72 hour period
  Other Names: advil
  Arms: Tx 2: ibuprofen and education; Tx 3: ibuprofen/acetaminophen/education

SUMMARY:
Concussions and headache are a significant problem for children and athletes. While headache generally resolves within 7-10 days; a significant proportion of children, 72-93% experience prolonged headache as a symptom of Post Concussion Syndrome (PCS). The prevailing clinical view is that mild head injuries resolve with little chance of complications. However, the reality is quite different. Concussion in children presents with a range of severity and results in both short and long-term physical, cognitive, emotional and behavioural sequelae known as PCS with varying times to resolution. To date there are no specific treatments for headache pain related to concussion. Physical and cognitive rest is the mainstay of initial concussion management.

The number of children presenting to ED's with a history of concussion and headache is increasing. Presently there are no evidence based guidelines available to guide the medical team to effectively and consistently manage their headache. Our present standard of care is based on the CANCHILD concussion guidelines outlining the child's return to school and activity. Yet, our present standard of treatment is compromised and somewhat counterproductive if we are not treating the child's headache pain.

Our pilot study ' An Open Label Randomized Control Pilot Study Examining Treatment of Headache In The Post-Concussive Youth' showed that routine administration of oral analgesia improves the child's headache symptoms and helps with school re-entry one week post injury, compared to a standard care group defined as non routine administration of pain medications.

DETAILED DESCRIPTION:
Objective Post Injury concussion and headache are problematic for children after mild traumatic brain injuries. There are no evidence based guidelines for the management of acute post concussive headache. The objectives of this study were to assess the efficacy of routine administration of analgesia on concussion headache and classify headaches using the IHS criteria.

Method A 4 arm open label pilot RCT study was conducted. The treatment arms were: (i) acetaminophen,(ii) ibuprofen, (iii) acetaminophen and ibuprofen and (iv) a standard control group. Eight to eighteen year olds presenting to emergency with headache 24-48 hours after their first concussion were recruited consecutively and sequentially randomized. Demographic data was collected, headache survey administered and standard concussion education given. Headaches were diarized over one week capturing the (i) number of headaches, (ii) headache days,(iii) headache intensity and (iv) return to school.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with a first time concussion
* english speaking
* presenting to Emergency with headache 24-48 hours post concussion
* normal Glascow Coma Scale
* 8-18 years of age

Exclusion Criteria

* postive findings on CT scan
* patient with cervical injury
* history of multiple concussions
* positive neurology

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina m Petrelli, PhD, Principal Investigator — McMaster Children's Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Youth presenting to pediatric tertiary centre ED within 48 hours of concussive event and having headache.
Groups:
- tx 1: Acetaminophen and Education: Patient took routinely acetaminophen every 4 hours when awake for a 72 hour period and documented their headaches for a week.
  Patient and family received standard education on concussion management in the Emergency department.
  Acetaminophen: routine administration of medication for a 72 hour period
- Tx 2: Ibuprofen and Education: Patient took routinely ibuprofen every 6 hours when awake for a 72 hour period and documented their headaches for a week.
  Patient and family received standard education on concussion management in the Emergency department.
  Ibuprofen: routine administration of medication for a 72 hour period
- Tx 3: Ibuprofen/Acetaminophen/Education: Patient took routinely ibuprofen (Q6H) and acetaminophen (Q4H) for when awake for 72 hours post concussion and documented their headaches for a week.
  Patient and family received standard education on concussion management in the Emergency Department.
  Acetaminophen: routine administration of medication for a 72 hour period
  Ibuprofen: routine administration of medication for a 72 hour period
Period: Overall Study
Arm/Group | tx 1: Acetaminophen and Education | Tx 2: Ibuprofen and Education | Tx 3: Ibuprofen/Acetaminophen/Education | Tx 4: no Routine Meds and Education
Started | 20 | 20 | 20 | 20
Completed | 19 | 20 | 20 | 20
Not Completed | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | tx 1: Acetaminophen and Education | Tx 2: Ibuprofen and Education | Tx 3: Ibuprofen/Acetaminophen/Education | Tx 4: no Routine Meds and Education | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (2.2) | 13.0 (2.6) | 12.3 (3.0) | 12.3 (2.4) | 13.1 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 8 | 9 | 40
  Male | 11 | 6 | 12 | 11 | 40
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 20 | 20 | 20 | 80
mechanism of injury [Number; unit: participants]
  fall | 3 | 6 | 4 | 5 | 18
  sports | 12 | 12 | 13 | 12 | 49
  motor vehicle accident | 2 | 0 | 0 | 1 | 3
  assault | 1 | 2 | 0 | 0 | 3
  other | 2 | 0 | 3 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Headache Days
Description: study participants completed a one week diary at home stating if they had headaches.
Time Frame: one week
Measure: Mean (Full Range); unit: number of headache days
Arm/Group | tx 1: Acetaminophen and Education | Tx 2: Ibuprofen and Education | Tx 3: Ibuprofen/Acetaminophen/Education | Tx 4: no Routine Meds and Education
Number analyzed (Participants) | 19 | 20 | 20 | 20
number of headache days | 4 [2 to 5] | 3 [3 to 4] | 3 [2 to 4] | 4 [4 to 6]

2. Secondary Outcome: Percentage of Study Participants That Returned to School at One Week Post Concussion
Description: patients/family were asked if the child returned to school one week after their injury
Time Frame: one week
Measure: Number; unit: percentage of participants
Arm/Group | tx 1: Acetaminophen and Education | Tx 2: Ibuprofen and Education | Tx 3: Ibuprofen/Acetaminophen/Education | Tx 4: no Routine Meds and Education
Number analyzed (Participants) | 19 | 20 | 20 | 20
percentage of participants | 33 | 61 | 79 | 21

3. Other Pre Specified Outcome: Headache Intensity Per Day for One Week
Description: The Numerical Rating Scale (NRS) will be used to capture the intensity of the headache experience. The NRS was initially developed for acute post procedural pain and is now a common measure for headache and disease related pain with well established reliability and validity as a self report measure in this age group. Children meeting the inclusion criteria also meet the criteria for self report. The numerical rating scale includes indicators from 0 to 10 with 0 being the 'no pain' and 10 being 'the worst pain ever'. The child when diarizing the headaches will report a pain intensity score for each headache type in their one week headache diary. Study participants and their parent will be given instruction regarding reporting the headache instruction. The headache intensity scores were averaged for the day per participant.
Time Frame: one week
Measure: Median (Full Range); unit: units on a scale
Arm/Group | tx 1: Acetaminophen and Education | Tx 2: Ibuprofen and Education | Tx 3: Ibuprofen/Acetaminophen/Education | Tx 4: no Routine Meds and Education
Number analyzed (Participants) | 19 | 20 | 20 | 20
units on a scale
  day one n=19, n=20, n= 20, n=20 | 8 [6 to 9] | 8 [6 to 9] | 7 [4 to 8] | 8 [6 to 9]
  day two n=19, n=20, n=20, n=20 | 6 [5 to 7] | 6 [4 to 6] | 5 [2 to 6] | 8 [6 to 9]
  day 3 n=19, n= 20, n=20, n=20 | 5 [4 to 6] | 4 [3 to 5] | 3 [2 to 4] | 6 [4 to 8]
  day 4 n=19, n=18, n=4, n=20 | 5 [3 to 6] | 3 [2 to 4] | 2.5 [2 to 3] | 6 [4 to 7]
  day five n=18, n=3, n=0, n=20 | 4 [3 to 6] | 3 [2 to 3] | NA [NA to NA] — no headaches reported | 5 [5 to 7]
  day 6 n=12, n=0, n=0, n=20, | 4 [3 to 5] | NA [NA to NA] — no headaches reported | NA [NA to NA] — no headaches reported | 5 [4 to 7]
  day 7 n=4, n=0, n=0, n=18 | 3.5 [3 to 6] | NA [NA to NA] — no headaches reported | NA [NA to NA] — no headaches reported | 5 [3 to 6]

4. Other Pre Specified Outcome: Number of Headaches a Day
Description: the patient family were given a headache diary and instruction to document the number of headaches they have a day for a one week period.
Time Frame: one week
Measure: Median (Full Range); unit: headaches per day
Arm/Group | tx 1: Acetaminophen and Education | Tx 2: Ibuprofen and Education | Tx 3: Ibuprofen/Acetaminophen/Education | Tx 4: no Routine Meds and Education
Number analyzed (Participants) | 19 | 20 | 20 | 20
headaches per day
  day one n=19, n=20, n= 20, n=20 | 4 [2 to 5] | 3 [3 to 4] | 3 [2 to 4] | 4 [4 to 6]
  day two n=19, n=20, n=20, n=20 | 4 [3 to 4] | 3 [3 to 4] | 2 [2 to 4] | 4 [3 to 5]
  day 3 n=19, n= 20, n=20, n=20 | 3 [2 to 4] | 3 [2 to 3] | 2 [1 to 3] | 4 [3 to 5]
  day 4 n=19, n=18, n=4, n=20 | 3 [2 to 4] | 2 [1 to 3] | 1 [1 to 1] | 4 [3 to 5]
  day four n=18, n=3, n=0, n=20 | 3 [1 to 4] | 1 [1 to 1] | NA [NA to NA] — no headaches reported | 4 [3 to 4]
  day 6 n=12, n=0, n=0, n=20, | 2 [1 to 3] | NA [NA to NA] — no headaches reported | NA [NA to NA] — no headaches reported | 3 [1 to 5]
  day 7 n=4, n=0, n=0, n=18 | 1 [1 to 1] | NA [NA to NA] — no headaches reported | NA [NA to NA] — no headaches reported | 3 [1 to 4]

ADVERSE EVENTS:
Description: serious and other adverse events were not collected.
Arm/Group | tx 1: Acetaminophen and Education | Tx 2: Ibuprofen and Education | Tx 3: Ibuprofen/Acetaminophen/Education | Tx 4: no Routine Meds and Education
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
open label study, not blinded pilot study, no sample size calculation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No